CLINICAL TRIAL: NCT06543459
Title: A Single-center, Randomized, Double-blind, Single Oral Dose, Placebo-controlled Study to Evaluate the Effect of MY008211A Tablets on QTc Interval in Healthy Chinese Adult Subjects
Brief Title: To Evaluate the Effect of Single Oral Dose of MY008211A Tablets on QTc Interval in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MY008211-1-07
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A, Sequence 1, Dose 1 (Experimental): Participants randomized to receive MY008211A tablets or placebo on Day 1.
  Interventions: Drug: MY008211A tablets
- Group A, Sequence 2, Dose 2 (Experimental): Participants randomized to receive MY008211A tablets or placebo on Day 7.
  Interventions: Drug: MY008211A tablets
- Group B, Sequence 1, Dose 1 (Placebo Comparator): Participants randomized to receive MY008211A tablets or placebo on Day 1.
  Interventions: Drug: Placebo
- Group B, Sequence 2, Dose 2 (Placebo Comparator): Participants randomized to receive MY008211A tablets or placebo on Day 7.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MY008211A tablets — Subjects of Group A receive MY008211A tablets on Day 1 of both Sequence, wash-out period is 6 Days at least.
  Arms: Group A, Sequence 1, Dose 1; Group A, Sequence 2, Dose 2
Drug: Placebo — Subjects of Group A receive placebo tablets on Day 1 of both Sequence, wash-out period is 6 Days at least.
  Arms: Group B, Sequence 1, Dose 1; Group B, Sequence 2, Dose 2

SUMMARY:
A Concentration-QT Interval Correction (C-QTc) study of MY008211A Tablets in Healthy Subjects

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, single oral dose, two groups, placebo-controlled study with 2 dose sequences preset

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers must be fully informed of this study and the content, process of the study and possible adverse events related to experimental drug will be fully understood, and voluntarily signed a written Informed Consent Form (ICF);
2. 18≤ age ≤ 45 years old, male or female Chinese adult volunteers;
3. Body weight: ≥50 kg for male, ≥45 kg for female; body mass index (BMI): 19.0-26.0 kg/m2 (inclusive) at screening;
4. Volunteers should be able to communicate well with the investigator, understand and comply with the requirements of the study.

Exclusion Criteria:

1. The investigator judges that there are other disease or medical conditions that are clinical significant or may prevent the volunteer from following the study protocol and completing the study, abnormal including but not limited to central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematological system, immune system, mental system, endocrine and metabolic system;
2. Volunteers with chronic or active gastrointestinal diseases such as esophageal disease, gastritis, gastric ulcer, enteritis, active gastrointestinal bleeding, or gastrointestinal surgery within the past three years and judged by the investigator to have clinical significance at present;
3. Volunteers with torsades de pointes (TDP) or other risk factors for malignant arrhythmias, or short QT syndrome, long QT syndrome, sudden unexplained death or drowning in youth (≤ 40 years old), or a family history of a first-degree relative (i.e., biological parent, sibling, or child) of sudden infant death syndrome, or other heart disease that the investigators determined was not suitable for inclusion;
4. Volunteers with hyperkalemia, hypokalemia, hypermagnesia, hypomagnesemia, hypercalcemia or hypocalcemia and judged by the investigator to have clinical significance;
5. History of known or suspected immunodeficiency (e.g., history of frequent recurrent infections), inherited or acquired complement deficiency；
6. Volunteers who underwent surgery within 6 months pre-dose, which judged by the investigator to affect the absorption, distribution, metabolism, and excretion of the experimental drug(e.g. cholecystectomy, except appendicitis surgery); Surgical procedures within 4 weeks pre-dose or planned to undergo a surgical procedure during the trial;
7. Volunteers who had a clear history of capsular microbial infection within 6 months before screening; Including but not limited to: Streptococcus pneumoniae, Bacillus anthracis, Salmonella, Salmonella typhi, Klebsiella pneumoniae, Pseudomonas aeruginosa, Bacteroides fragilis, Neisseria meningitidis, Haemophilus influenzae, Legionella pneumophila infection history;
8. Volunteers with previous or current history of TB infection or with positive lymphobacteria culture + interferon test；
9. Active systemic bacterial, viral, or fungal infection within 14 days pre-dose;
10. Fever (≥ 38 ℃) within 7 days pre-dose;
11. Volunteers with a history of clinically significant drug allergy or allergic disease (such as asthma, urticaria, eczematous dermatitis, etc.), or a possible or clear allergy to the experimental drug (including similar drugs) or any excipients thereof as judged by the investigator;
12. Volunteers with clinical significant examination abnormalities which judged by the investigator such as vital signs, physical examination, routine laboratory tests (can reviewable, including: blood routine, reticulocyte count, procalcitonin + myoglobin, blood biochemical + hypersensitive C-reactive protein, urine routine, coagulation function + plasma D-Dimer determination), chest X-ray, abdominal ultrasound at screening or baseline；
13. Volunteers with 12-ECG examination and reviewable result such as QTcF≥450 ms or PR interval ≥200ms or QRS wave complex ≥120ms or clinical significant abnormality ECG which judged by the investigator at screening or baseline or pre-dose；
14. Volunteers who administrated any other clinical study drug or enrolled in any Interventional clinical trial within 3 months before screening；
15. Volunteers who donated blood or lost blood (≥ 400mL) within 3 months pre-dose, received a blood transfusion or use of blood products within 4 weeks pre-dose, or intended to donate blood or blood components during or within 3 months after study;
16. Volunteers who had taken any medicine or OTC medicine or Chinese herbal medicine or food supplement (including vitamins, health foods, etc.) other non-drug therapeutic factors that affect drug absorption, distribution, metabolism and excretion;
17. Volunteers who received a vaccine or live attenuated vaccine within 14 days pre-dose, or who plan to receive a vaccine during the study;
18. Volunteers with difficulty in blood collection or cannot tolerate intravenous puncture;
19. Volunteers with a history of drug use or substance abuse or with positive urine drug abuse screening test;
20. Volunteers with any positive result of virological test;
21. Volunteers who drink more than 14 units a week (one unit is defined as 360mL of beer or 45mL of liquor or 150mL of wine) within 3 months before screening or with positive result of alcohol breath test or unwillingness to stop drinking alcohol or any alcohol-based product during the study；
22. Volunteers who smoke more than 5 cigarettes per day(or use a significant amount of nicotine products) within 3 months before screening or will be unable to stop using any tobacco products during the study or with positive result of urine nicotine test；
23. Volunteers who habitual consumption of grapefruit juice or excessive amounts of tea, coffee and/or caffeinated beverages and will be unable to stop use during the study, or consume any food or drink containing chocolate, caffeine, or rich in xanthines within 48h pre-dose；
24. Volunteers who have special requirements for diet and cannot abide by the uniform diet；
25. Volunteers (or their partners) who plan to be pregnant or donate sperm or eggs during the study to 3 months after the end of the study, or who are unwilling to take one or more non-drug contraceptive measures (such as complete abstinence, condoms, contraceptive rings, surgical sterilization, etc.);
26. Volunteers of pregnant or lactating women; or having unprotected sex within 2 weeks pre-dose; or oral contraceptive use within 30 days or long-acting estrogen or progestin injectable or implant use within 6 months pre-dose; or with positive blood pregnancy test pre-dose;
27. Volunteers have other reasons for not fit for participating in the study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-09-27 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
ΔΔQTcF (Using Fridericia Formula as the Primary Method for QT Interval Correction) | up to 2 weeks
  Placebo-corrected, baseline-adjusted QTc interval of prodrug and active metabolite (if necessary)

SECONDARY OUTCOMES:
Cmax (Maximum plasma concentration) | up to 2 weeks
  Cmax of prodrug and active metabolite (if necessary)
Tmax (Time to maximum plasma concentration) | up to 2 weeks
  Tmax of prodrug and active metabolite (if necessary)
t1/2 (Terminal elimination half-life time) | up to 2 weeks
  t1/2 of prodrug and active metabolite (if necessary)
AUC0-t (Area under the plasma concentration-time curve from time 0 to the collection time t with the last measurable plasma concentration) | up to 2 weeks
  AUC0-t of prodrug and active metabolite (if necessary)
AUC0-∞ (Area under the plasma concentration-time curve extrapolated from time 0 to infinity) | up to 2 weeks
  AUC0-∞ of prodrug and active metabolite (if necessary)
CL/F (Apparent clearance) | up to 2 weeks
  CL/F of prodrug and active metabolite (if necessary)
Vz/F (Apparent volume of distribution) | up to 2 weeks
  Vz/F of prodrug and active metabolite (if necessary)
The incidence and severity of adverse events to assess safety and tolerability | up to 3 weeks
  such as laboratory abnormalities
Other Electrocardiogram (ECG) parameters | up to 2 weeks
  Such as T-wave morphology or absence, U-wave presence and absence, HR, RR interval, PR interval, QRS wave complex

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Li, PhD, Principal Investigator — PI
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Trade secrets